CLINICAL TRIAL: NCT05813535
Title: Sodium Bicarb Locks in Intestinal Failure
Brief Title: 8.4% Sodium Bicarbonate Locks in Intestinal Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riad Rahhal (Other)
Responsible Party: Sponsor-Investigator, Riad Rahhal, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202205087
Record Dates: First submitted 2023-03-20; First posted 2023-04-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Intestinal Failure; CRBSI - Catheter Related Bloodstream Infection
MeSH Terms: conditions — Intestinal Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baseline (Other): Patient on heparin locks when off venous nutrition
  Interventions: Drug: Sodium bicarb lock

INTERVENTIONS:
Drug: Sodium bicarb lock — 8.4% sodium bicarb locks when off venous nutrition

SUMMARY:
We plan to include children with intestinal failure, a condition where the gut is not functioning properly, leading these children to need central venous catheters (line that goes through the skin into the blood stream) for nutritional support and hydration. Such patients have a very high risk for catheter infection. The study will include placing an agent (sodium bicarbonate) into the central catheter when the catheter is not in use. This is referred to as a lock. The lock would be used daily and removed when patients start their nutritional support and hydration through the catheter.

DETAILED DESCRIPTION:
Children with intestinal failure who rely on a silicone based central venous catheter for parenteral nutrition to provide nutritional support and hydration will be invited to participate in this study. The intervention will offer use of a specific catheter lock solution (8.4% sodium bicarbonate) when the catheter is not in use. This includes daily lock use with removal of the lock at end of dwell time.

ELIGIBILITY:
Inclusion Criteria:

* Subject fulfills diagnosis of intestinal failure with a central venous catheter in place used daily on outpatient basis for intravenous nutrition and /or intravenous hydration
* Subject is less than 18 years of age at the time of study entry
* Subject with history of at least 1 documented catheter related blood stream infection (verified by blood culture)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of catheter related bloodstream infections | Through study completion, an average of 1 year
  Number of infections per 1000 catheter days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States